CLINICAL TRIAL: NCT00003677
Title: Phase II Study of Dolastatin 10 (NSC# 376128) Administered Intravenously Every 21 Days to Patients With Metastatic Pancreatic Adenocarcinoma
Brief Title: Dolastatin 10 in Treating Patients With Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM98-071; P30CA016672 (NIH); U01CA070172 (NIH); U01CA063187 (NIH); MDA-DM-98071 (Other: UT MD Anderson Cancer Center); NCI-T98-0028; CDR0000066778 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-07-22 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Pancreatic Cancer
Keywords: recurrent pancreatic cancer; adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — dolastatin 10

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dolastatin 10 (Experimental): Dolastatin 10 IV bolus once every 21 days.
  Interventions: Drug: Dolastatin 10

INTERVENTIONS:
Drug: Dolastatin 10 — IV bolus once every 21 days.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of dolastatin 10 in treating patients who have metastatic pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the antitumor activity of dolastatin 10 in patients with metastatic adenocarcinoma of the pancreas. II. Evaluate the qualitative and quantitative toxic effects of this therapy in these patients. III. Investigate the clinical pharmacology of this treatment.

OUTLINE: This is an open label, multicenter study. Patients receive dolastatin 10 IV bolus once every 21 days. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months until death.

PROJECTED ACCRUAL: This study will accrue 12-37 patients within 18.5 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed metastatic adenocarcinoma of the pancreas Bidimensionally measurable lesions with sentinel lesions outside field of any prior radiation therapy No brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Zubrod 0-1 Life expectancy: At least 12 weeks Hematopoietic: Absolute granulocyte count at least 1500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL Renal: Creatinine no greater than 1.5 mg/dL Cardiovascular: No active congestive heart failure No uncontrolled angina At least 6 months since prior myocardial infarction No uncontrolled hypertension Other: Not pregnant or nursing Fertile patients must use effective contraception No concurrent serious infection At least 5 years since prior malignancy except the following: Nonmelanoma skin cancer Carcinoma in situ of the cervix No overt psychosis or mental disability

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent biologic therapy Chemotherapy: No prior chemotherapy for metastatic disease At least 6 months since prior adjuvant chemotherapy No concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics At least 6 months since prior adjuvant chemoradiation to disease At least 2 weeks since prior radiotherapy and recovered No concurrent radiotherapy Surgery: At least 4 weeks since prior surgery and recovered No concurrent surgery Other: At least 4 weeks since prior investigational drug (including analgesics or antiemetics) No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 1999-02-01 (Actual); Primary Completion 2002-01-16 (Actual); Study Completion 2002-01-16 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Toxicity | Every 3 months
  Toxic effects of dolastatin 10 therapy in patients with metastatic adenocarcinoma of the pancreas used to assess antitumor activity.

CONTACTS AND LOCATIONS:
Overall Officials: Hedy L. Kindler, MD, Study Chair — University of Chicago
Locations (2):
- United States (2):
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - University of Texas - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org